CLINICAL TRIAL: NCT05843032
Title: 3D Ultrasound in the Assessment of Resection Margins During Surgery for Squamous Cell Carcinoma of the Tongue: a Comparison With Clinical Evaluation, MRI, and Histopathology
Brief Title: 3D Ultrasound, Specimen Examination by Surgeon, and MRI in Surgical Margin Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Fatemeh Makouei, Biomedical Engineer, PhD, Assistant professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21017915
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Squamous Cell Carcinoma; Tongue SCC; Head and Neck Cancer
Keywords: Ultrasound; 3D ultrasound; Ultrasonography; Three dimensional imaging; cancer diagnosis; surgical margin assessment; magnetic resonance imaging; MRI; ex-vivo surgical specimen imaging; squamous cell carcinoma; histopathology; SCC; oral cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Mouth Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tongue tumor resection (Experimental)
  Interventions: Diagnostic Test: 3D ultrasound, MRI, resected specimen examination by surgeon

INTERVENTIONS:
Diagnostic Test: 3D ultrasound, MRI, resected specimen examination by surgeon — 3D ultrasound and MR scanning of the resected tongue tumor will be performed. The resected surgical specimen will also be examined by the surgeon to assess the margins. The accuracy of the margin assessment by 3D ultrasound, MRI, and surgeon examination will be evaluated by correlating the results to the final histopathology findings.

SUMMARY:
In the current protocol, application of 3D ex-vivo ultrasound, MRI, and clinical evaluation (palpation and examination) by the surgeon is proposed to analyze the margin status in tongue squamous cell carcinoma and correlate the results to the histopathology findings.

DETAILED DESCRIPTION:
Cancer surgery is the primary treatment in the early stages of tongue squamous cell carcinoma (SCC), and the goal is the complete resection of the tumor with an adequate margin of healthy tissue around to ensure proper cancer removal. Inadequate margins lead to a high risk of local cancer recurrence and the patient will need re-surgery or adjuvant therapies. Ex-vivo imaging of the resected surgical specimen has been suggested to provide information for margin assessment and thus improve cancer surgery. In this manuscript, a protocol to investigate the clinical benefit of three-dimensional (3D) ultrasound imaging of the surgical margins and comparing the results to magnetic resonance imaging (MRI) and the clinical examination of the surgical specimen by surgeon (palpation to inspect the resected tissue) has been designed. Tumor segmentation and margin measurement (Anterior towards apex of tongue, posterior towards base of tongue, medial towards back of tongue, lateral towards floor of mouth, and profound/deep margins) will be performed by head and neck surgeons on 3D ultrasound images and by two consultant radiologists on MRI of the ex-vivo specimen. Accuracy of each method will be evaluated by computing the proportion of correctly classified margins (positive, close, and free) by each technique with respect to the gold standard histopathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven oral tongue squamous cell carcinoma scheduled for surgical treatment
* T1-T3 staging on cross-sectional imaging

Exclusion Criteria:

* T4 staging
* Unable to understand the verbal or written information
* Prior radiotherapy treatment of oral cavity cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the 3D ultrasound and MRI compared to the conventional method in measurements of the surgical margins in the resected tongue SCC specimens. | 2 weeks
Diagnostic accuracy - number of margins correctly classified as free (> 5 mm), close (1- 5 mm) or positive (<1 mm) margin by 3D ultrasound and MRI using histopathology findings as the reference | 2 weeks

SECONDARY OUTCOMES:
Number of cases requiring adjuvant treatments (surgery or chemo/radiotherapy) | 2 weeks
Shrinkage of the surgical specimen due to formalin fixation based on the specimen volume measurements on 3D ultrasound images before and after formalin fixation | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Available for 5 years

REFERENCES:
- [Background] Chinn SB, Myers JN. Oral Cavity Carcinoma: Current Management, Controversies, and Future Directions. J Clin Oncol. 2015 Oct 10;33(29):3269-76. doi: 10.1200/JCO.2015.61.2929. Epub 2015 Sep 8. PMID 26351335
- [Background] Pagedar NA. Better Visualization of Oral Cancer Margins-A Struggle of Cancer and Technology. JAMA Otolaryngol Head Neck Surg. 2020 Dec 1;146(12):1156-1157. doi: 10.1001/jamaoto.2020.3262. No abstract available. PMID 33030524
- [Background] Schmidt Jensen J, Jakobsen KK, Mirian C, Christensen JT, Schneider K, Nahavandipour A, Wingstrand VL, Wessel I, Tvedskov JF, Frisch T, Christensen A, Specht L, Andersen E, Lelkaitis G, Gronhoj C, von Buchwald C. The Copenhagen Oral Cavity Squamous Cell Carcinoma database: protocol and report on establishing a comprehensive oral cavity cancer database. Clin Epidemiol. 2019 Aug 19;11:733-741. doi: 10.2147/CLEP.S215399. eCollection 2019. PMID 31695503
- [Background] de Koning KJ, Koppes SA, de Bree R, Dankbaar JW, Willems SM, van Es RJJ, Noorlag R. Feasibility study of ultrasound-guided resection of tongue cancer with immediate specimen examination to improve margin control - Comparison with conventional treatment. Oral Oncol. 2021 May;116:105249. doi: 10.1016/j.oraloncology.2021.105249. Epub 2021 Mar 26. PMID 33774501
- [Background] Narayana HM, Panda NK, Mann SB, Katariya S, Vasishta RK. Ultrasound versus physical examination in staging carcinoma of the mobile tongue. J Laryngol Otol. 1996 Jan;110(1):43-7. doi: 10.1017/s0022215100132682. PMID 8745780
- [Background] Klein Nulent TJW, Noorlag R, Van Cann EM, Pameijer FA, Willems SM, Yesuratnam A, Rosenberg AJWP, de Bree R, van Es RJJ. Intraoral ultrasonography to measure tumor thickness of oral cancer: A systematic review and meta-analysis. Oral Oncol. 2018 Feb;77:29-36. doi: 10.1016/j.oraloncology.2017.12.007. Epub 2017 Dec 18. PMID 29362123
- [Background] Tarabichi O, Bulbul MG, Kanumuri VV, Faquin WC, Juliano AF, Cunnane ME, Varvares MA. Utility of intraoral ultrasound in managing oral tongue squamous cell carcinoma: Systematic review. Laryngoscope. 2019 Mar;129(3):662-670. doi: 10.1002/lary.27403. Epub 2018 Aug 27. PMID 30151976
- [Background] de Koning KJ, van Es RJJ, Klijn RJ, Breimer GE, Willem Dankbaar J, Braunius WW, van Cann EM, Dieleman FJ, Rijken JA, Tijink BM, de Bree R, Noorlag R. Application and accuracy of ultrasound-guided resections of tongue cancer. Oral Oncol. 2022 Oct;133:106023. doi: 10.1016/j.oraloncology.2022.106023. Epub 2022 Jul 25. PMID 35901543
- [Background] Makouei F, Ewertsen C, Agander TK, Olesen MV, Pakkenberg B, Todsen T. 3D Ultrasound versus Computed Tomography for Tumor Volume Measurement Compared to Gross Pathology-A Pilot Study on an Animal Model. J Imaging. 2022 Dec 19;8(12):329. doi: 10.3390/jimaging8120329. PMID 36547494